CLINICAL TRIAL: NCT06514183
Title: Long Term Post-treatment Follow-up After End of Study (>15 Months) of Clinical Trial Participants Enrolled in DNDi-FOSR-04-MYC
Brief Title: Eumycetoma Long-term Post-Treatment Follow-Up Study
Status: Terminated | Type: Observational
Why Stopped: Due to the socio-political sutuation in Sudan affecting patient follow-up
Sponsor: Drugs for Neglected Diseases (Other)
Collaborators: Soba University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: DNDi-FOSR-05-MYC
Record Dates: First submitted 2023-03-22; First posted 2024-07-23 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Eumycetoma
Keywords: Mycetoma; Madura foot; Madurella mycetomatis
MeSH Terms: conditions — Mycetoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Biopsy of masses on the infected sites and serum samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Clinical diagnosis of recurrence — Clinical diagnosis of recurrence

SUMMARY:
To assess the long-term recurrence rate of eumycetoma in clinical trial participants treated in the phase II DNDi-FOSR-04-MYC clinical trial.

DETAILED DESCRIPTION:
The purpose of the long-term post treatment follow-up study is to collect data on recurrence of eumycetoma lesions in participants who previously participated in: A randomized, double blind phase II proof-of-concept superiority trial of fosravuconazole 200 mg or 300 mg weekly dose versus itraconazole 400 mg daily, all three arms in combination with surgery, in participants with eumycetoma in Sudan (DNDi-FOSR-04-MYC).

These data will provide additional information on recurrences after end of study (>15 months) of the parent clinical trial (DNDi-FOSR-04-MYC). The study is observational, since there is no intervention in this protocol, but assesses the outcome of the intervention of the parent trial.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical trial participants who were previously enrolled and received investigational product (fosravuconazole) or standard of care treatment (itraconazole) in the DNDi-FOSR-04-MYC clinical trial.
2. In trial DNDi-FOSR-04-MYC had no recurrence of eumycetoma lesion before month 15.
3. Able and willing to give written informed consent for participation in this study, prior to performance of any study procedures.

Exclusion Criteria:

1. Any condition that, in the opinion of the Principal Investigator or designee, would preclude provision of informed consent or interfere with achieving the study objectives.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will consist of the clinical trial participants that were recruited in the RCT trial DNDi-FOSR-04-MYC. The RCT had enrolled 104 clinical trial participants with 29 having recurrence before month 15. Therefore, the long-term post-treatment follow-up assessment will target 75 participants that had no recurrence indicated at end of study or who had not completed the study i.e., those who had been regarded as lost to follow up but may now be available.
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2023-01-26 (Actual); Primary Completion 2023-06-26 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
To assess recurrence of eumycetoma lesions up to 5 years after end of treatment in participants previously treated with fosravuconazole 200 mg or 300 mg weekly or itraconazole 400 mg daily in study DNDi-FOSR-04-MYC | 6 years
  Population: Participants in trial DNDi-FOSR-04-MYC who had no recurrence of eumycetoma lesion before month 15
  * Treatment: fosravuconazole 200 mg or 300 mg weekly or itraconazole 400 mg daily in study DNDi-FOSR-04-MYC
  * Variable: Time to recurrence of eumycetoma lesion (if lesion occurred) or time followed-up without lesion

SECONDARY OUTCOMES:
To determine efficacy of fosravuconazole 200 mg or 300 mg monotherapy vs. itraconazole monotherapy, after long term post-treatment follow-up | 15 months
  Population/Treatment/Variable/Intercurrent events: as for primary estimand Hazard ratios comparing a) risk of recurrence for fosravuconazole 200mg vs. itraconazole
To assess overall recurrence of eumycetoma lesions up to 5 years in participants treated with fosravuconazole 200 mg or 300 mg weekly or itraconazole 400 mg daily in study DNDi-FOSR-04-MYC | 6 years
  Population: Participants in trial DNDi-FOSR-04-MYC regardless of recurrence before Month 15.
  Treatment/Variable/Intercurrent events: as defined for the primary estimand
To describe the etiologic pathogen (subtype of fungus) after long term recurrence | 15 months
  Population: Participants with recurrence of eumycetoma within the current study Summary measure: Proportion of recurrences of each subtype
  * Treatment: as for primary estimand
  * Variable: Typing of fungus

CONTACTS AND LOCATIONS:
Overall Officials: Borna A Nyaoke, M.D, Study Director — Drugs for Neglected Diseases initiative
Locations (1):
- Mycetoma Research Center, Soba University Hospital, Khartoum, Sudan

IPD SHARING:
Plan to Share IPD: Yes
Through Drugs for Neglected Diseases Initiative (DNDi) and open data sharing platforms. The data may be obtained by sending a request to DNDi
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Currently available with no end date
Access Criteria: Must adhere to appropriate agreement or terms of use and contractual obligations which DNDi may have with its partners.
URL: http://dndi.org